CLINICAL TRIAL: NCT06561724
Title: The Application of Potential Biotechnologies to Develop Novel Probiotics Functional Food Products With High Viability for Modulating the Gut Microbiome Among Healthy and Under Stress Subiects
Brief Title: Diet Supplementation With Prebiotics to Improve Gut Health in Egyptian Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Collaborators: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7445052023
Record Dates: First submitted 2024-04-09; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-02

CONDITIONS: Microbial Colonization; Gut Microbiota
Keywords: Gut microbiome; Diarrhea; Irritable bowel syndrome; Inulin prebiotic; Metagenomic analysis; Fecal Secretory immunoglobulin A; Fecal short chain fatty acids
MeSH Terms: conditions — Communicable Diseases; Diarrhea; Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomized blind parallel three -arm randomized controlled trial (RCT). The RCT is double-blind, in which both the nutritionist and the volunteers are blinded to the actual biscuit allocated to the volunteer; i.e., neither the nutritionist in charge of distributing the biscuit nor the volunteer knows whether the volunteer has received prebiotic rich biscuit or placebo.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Biscuits includes maltodextrin (Active Comparator): Maltodextrin is a generally recognized as safe (GRAS) food additive. Functional maltodextrin biscuits were prepared by stacking the biscuits on the table, followed by dispensing of 2g maltodextrin. The biscuits were covered with another piece of biscuit and 1 g of honey was used as binder. The biscuits were packed in bags under vacuum and kept at 40C for the daily supply to the participants.
  Interventions: Dietary Supplement: Biscuits maltodextrin
- Biscuits includes prebiotics tartoufa inulin (Experimental): Prebiotics is the term for a dietary approach that tries to precisely control the composition and operation of the gut microbiota to promote health. Functional prebiotics biscuits were prepared by stacking the biscuits on the table, followed by dispensing of 2g tartoufa inulin. The biscuits were covered with another piece of biscuit and 1 g of honey was used as binder. The biscuits were packed in bags under vacuum and kept at 40C for the daily supply to the participants.
  Interventions: Dietary Supplement: Biscuits includes prebiotics tartoufa inulin
- Biscuits includes prebiotics chicory inulin (Experimental): Prebiotics is the term for a dietary approach that tries to precisely control the composition and operation of the gut microbiota to promote health. Functional prebiotics biscuits were prepared by stacking the biscuits on the table, followed by dispensing of 2g chicory inulin. The biscuits were covered with another piece of biscuit and 1 g of honey was used as binder. The biscuits were packed in bags under vacuum and kept at 40C for the daily supply to the participants.
  Interventions: Dietary Supplement: Biscuits includes prebiotics chicory inulin

INTERVENTIONS:
Dietary Supplement: Biscuits maltodextrin — Biscuits includes maltodextrin
  Arms: Biscuits includes maltodextrin
Dietary Supplement: Biscuits includes prebiotics tartoufa inulin — Biscuits prebiotics
  Arms: Biscuits includes prebiotics tartoufa inulin
Dietary Supplement: Biscuits includes prebiotics chicory inulin — Biscuits prebiotics
  Arms: Biscuits includes prebiotics chicory inulin

SUMMARY:
The study described herein seeks to assess the extent to which diet supplementation of young Egyptian children, one of the most vulnerable groups to the risk of diarrhea, with prebiotic fiber can improve their gut health.

DETAILED DESCRIPTION:
The gastrointestinal tract (GI) is an indispensable organ for any human. In addition to digesting and extracting nutrients from consumed foods, it also houses the largest community of human-associated microbes (called human gut microbiota), plays a role in immune system development and modulation, participates in water and electrolyte balancing, and excretes waste products. Because the human gut is constantly affected by external stimuli and foreign objects via food ingestion, it is not surprising that GI tract diseases, and especially diarrheal disease, are one of the most common causes of human illness. Diarrhea is especially prevalent at younger age, and indeed many young Egyptian children are vulnerable to develop such illness.

Healthy GI tract is the most densely populated human-associated microbial habitat and harbors a highly diverse microbial community. This gut microbiota functions as an essential organ in nutrition, immunity, and physiology of human hosts. Gut microbes are responsible for polysaccharide hydrolysis, vitamin production, immune system stimulation, and modulation of gut motility. While healthy gut microbiome provides protection of the human host against pathogen invasion, microbiota disbalance opens doors for the host to be colonized by intestinal pathogens including viruses, virulent bacteria, and parasites, which all can cause diarrhea. The burden of gut infections is high in Egypt, especially among young children. The vulnerability of these groups to gut infections has been linked previously to the level of hygiene and the integrity of intestinal barrier function, and can also be associated with the prevalence of pathogenic microbes in consumed foods such as poultry. The consumption of contaminated food and water, poor health knowledge, and ineffective infection control programs are contributing considerably to the persistence of enteric infections.

One of the approaches to reduce the prevalence of intestinal infections and resulting diarrhea is to improve overall gut health, by promoting the development of healthy gut microbiota and strengthening gut barrier function. Many dietary components can affect the composition and function of human gut microbiome. Among these, dietary fiber constitutes a variety of polysaccharides that are largely undigested and unabsorbed by humans (who lack enzymes required to break them), but are readily degraded by microbes in the large bowel. Fiber species that are selectively utilized by microbes and provide health benefits to the host are called prebiotics. These prebiotic fibers, such as inulin, selectively promote growth and expansion of beneficial members of our gut community, thus making it harder for pathogens to establish themselves in the gut. Fiber degradation by resident gut microbes also increases the levels of beneficial short chain fatty acids (SCFAs), which were shown to improve gut barrier function and reduce tissue inflammation.

ELIGIBILITY:
Inclusion Criteria:

• The inclusion criteria were children aged ≥3 and below 6 years and the ability of the child's mother to comply with the research protocol and to collect the biological materials at predetermined dates.

Exclusion Criteria:

* gastrointestinal diseases
* chronic diseases (such as type 1 diabetes)
* intake of antibiotics within the previous 3 months.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Fecal secretory immune globulin A (sIgA) | 2 months
  Fecal secretory s-IGA was assayed by the Chrom ELISA kit (Bio Vender research Diagnostics, Cat # RIC6100, Germany) and the instruction of the manufacturer was followed. Aliquots (80-120 mg) of the thawed fecal samples collected above at baseline and at the termination of the trial were suspended in 10-fold exes (15 m) shitoog a phspaste burier protered and entrifuged at 3o0 omn for s min. Tipes were simultaneously run in the ELISA and the concentration of s-IgA was read at 405 mm in ELISA reader against a standard curve and the results were expressed as mg faecal S-IgA per 100 gram stool.

SECONDARY OUTCOMES:
Fecal Short-chain fatty acids | 3 months
  The dry fecal sample was resuspended in 5ml 0.5 % ortho-phosphoric acid in the presence of 250 μl of the pure isobutyric acid as internal standard. Aliquots (60 μl) of the clear supernatant was aspirated and pipetted in a dry clean centrifuge tube containing 240 μl of 0.5% aqueous ortho-phosphoric acid, followed by the addition of 300 μl absolute butanol. Following vigorous shaking, the tubes were centrifuged and the clear supernatant was filtered through a Sartorius membrane filter of 0.25 microns. Aliquots (2 μl) were injected in Gas Chromatograph with a flame ionization detector (FID). The short-chain fatty acid concentrations were expressed in micromoles per gram of dry feces.
16s rRNA | 3 months
  Metagenomic analysis will be performed. Weighed aliquots (150 mg) of the thawed fecal samples were used for the genomic DNA extraction using the commercial fecal DNA Miniprep Zymo Research kit. The instruction of the manufacturer was followed. The concentration of the harvested DNA in the elute was determined by measuring the optical densities at 230 /260 nm using a nano spectrophotometer. The gnomic DNA is saved at -800C until metagenomic analysis. Standard protocols will be followed with the technical collaboration of Dr Oleg Paily.

CONTACTS AND LOCATIONS:
Overall Officials: Mosab Gad, PhD, Study Chair — National Research Centre, Egypt; Amr Elbahnasawy, PhD, Study Chair — National Research Centre, Egypt; Sahar Abdelaziz, PhD, Study Chair — National Research Centre, Egypt; Laila Hussein, PhD, Principal Investigator — National Research Centre, Egypt; Oleg Paliy, PhD, Principal Investigator — Wright State University, USA
Locations (1):
- Mosab Gad, Dokki, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared after publications
Time Frame: The data will be shared after publications
Access Criteria: Open data access

REFERENCES:
- [Background] Gad M, Elbahnasawy AS, Ramadan AA, Yamamah GAN, Hussein L. Dietary intervention with edible film-coated multistrain probiotic Lacticaseibacilli in nondairy food matrices significantly increased the recovery of fecal viable Lacticaseibacilli and improved the performance of several colonic biomarkers among slightly malnourished preschool children. Food Funct. 2024 Jan 22;15(2):977-991. doi: 10.1039/d3fo02829a. PMID 38179614
- [Background] Mohammad MA, Molloy A, Scott J, Hussein L. Plasma cobalamin and folate and their metabolic markers methylmalonic acid and total homocysteine among Egyptian children before and after nutritional supplementation with the probiotic bacteria Lactobacillus acidophilus in yoghurt matrix. Int J Food Sci Nutr. 2006 Nov-Dec;57(7-8):470-80. doi: 10.1080/09637480600968735. PMID 17162326
- [Background] Grimaldi R, Gibson GR, Vulevic J, Giallourou N, Castro-Mejia JL, Hansen LH, Leigh Gibson E, Nielsen DS, Costabile A. A prebiotic intervention study in children with autism spectrum disorders (ASDs). Microbiome. 2018 Aug 2;6(1):133. doi: 10.1186/s40168-018-0523-3. PMID 30071894